CLINICAL TRIAL: NCT01922193
Title: A Randomized, Assessor-blinded, Parallel Group, Multi-center, Non-inferiority Study Investigating the Efficacy and Safety of Highly Purified Urofollitropin for Injection Compared to Recombinant Human Follitropin Alfa for Injection in Controlled Ovarian Stimulation in Chinese Females Undergoing an Assisted Reproductive Technology (ART) Program
Brief Title: Evaluation of Efficacy and Safety of Highly Purified Urofollitropin in Chinese Females Undergoing an Assisted Reproductive Technology (ART) Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000089
Record Dates: First submitted 2013-07-24; First posted 2013-08-14 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Urofollitropin; follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Drug: Highly Purified Urofollitropin
- Control Group (Active Comparator)
  Interventions: Drug: Recombinant Human Follitropin Alfa

INTERVENTIONS:
Drug: Highly Purified Urofollitropin — for injection
  Other Names: Bravelle®
  Arms: Test Group
Drug: Recombinant Human Follitropin Alfa — for injection
  Other Names: Gonal-F®
  Arms: Control Group

SUMMARY:
Evaluate the efficacy and safety of of Highly Purified Urofollitropin for Injection Compared to Recombinant Human Follitropin Alfa for Injection in Chinese Females Undergoing an Assisted Reproductive Technology (ART) Program.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form, prior to screening evaluations
* In good physical and mental health
* Chinese Females between the ages of 20-39 years.
* Body mass index (BMI) is ≥ 18.5 and < 28 kg/m2
* Female diagnosed for at least one year (i.e., before screening) with tubal infertility, unexplained infertility, male factor infertility
* Regular menstrual cycles of 24-35 days (both inclusive), presumed to be ovulatory
* Documented evidence of at least one of the following within ninety (90) days prior to down regulation treatment:

  * mid-luteal phase serum progesterone level > 5ng/mL, or
  * late luteal phase endometrial biopsy with < 3 days lag, or
  * biphasic basal body temperature chart, or
  * mid-cycle urinary LH (Luteinizing hormone)surge
* Early follicular phase (day 2-3), serum levels of FSH within limits (1-12IU/L)(results obtained within 90 days prior to down regulation treatment)
* LH, PRL (prolactin), E2 (Estradiol), P (progesterone), total testosterone levels within normal range for the clinical laboratory or considered not clinically significant by the investigator (results obtained within 90 days prior to down regulation treatment)
* TSH (thyrotropin) levels within normal limits for the clinical laboratory or considered not clinically significant by the investigator, or secondary to exogenous thyroid medication (results obtained within 90 days prior to down regulation treatment)
* Negative serum Human Immunodeficiency Virus (HIV) antibody, and TPPA (Treponema Pallidum antibodies)/ RPR (Rapid Plasma Reagin) tests (results obtained within 90 days prior to down regulation treatment)
* Early follicular phase total antral follicle (diameter 2-10 mm) count ≥ 6 and ≤ 25 for both ovaries combined (results obtained within 3 months prior to down regulation treatment)
* Transvaginal ultrasound documenting presence and adequate visualisation of both ovaries, uterus and adnexa without evidence of significant abnormality (e.g.no endometrioma greater than 3 cm, no ovarian cysts > 35 mm or enlarged ovaries which would contraindicate the use of down regulation treatment, no hydrosalpinx) within ninety (90) days prior to down regulation treatment
* Hysterosalpingography, hysteroscopy, saline infusion sonography or transvaginal ultrasound documenting a uterus consistent with expected normal function (e.g.no evidence of clinically interfering uterine fibroids defined as submucous or intramural fibroids larger than 3 cm in diameter, no polyps and no congenital structural abnormalities which are incompatible with pregnancy) within 1 year prior to down regulation treatment. This also includes women who have been diagnosed with any of the above medical conditions but have had them surgically corrected.
* A minimum of one cycle without treatment with fertility modifiers (e.g., oral contraceptives) during the last menstrual cycle before down regulation treatment
* Willing to accept a maximum of two embryos transferred in the fresh cycle
* Willing to use an adequate barrier method of contraception or refrain from intercourse from 2 weeks before start of down regulation and throughout the down regulation period

Exclusion Criteria:

* Any pregnancy within last three (3) months prior to screening
* Known past or current thrombophlebitis or thromboembolism including venous thrombosis disease and active or recent arterial thrombosis disease
* Three or more controlled ovarian stimulation cycles for IVF/ICSI (In vitro fertilization/Intracytoplasmic sperm injection) prior to screening
* Previous IVF or ART failure related to a sperm/fertilization problem which resulted in unsuccessful fertilization and no related medical conditions improved
* Known history of poor ovarian response in a previous controlled ovarian stimulation cycle for IVF/ICSI
* Known history of excessive ovarian response in a previous controlled ovarian stimulation cycle for IVF/ICSI
* Known severe OHSS (Ovarian hyperstimulating syndrome) in a previous controlled ovarian stimulation cycle.
* Known history of polycystic ovary disease (PCOD) associated with anovulation
* Known endometriosis
* Known abnormal results of cervical examination of clinical significance obtained within 1 year prior to screening
* Abnormal vaginal bleeding of undetermined origin
* Known tumors of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus
* Known current active pelvic inflammatory disease
* Known history of recurrent miscarriage
* Known malformations of the sexual organs incompatible with pregnancy
* According to the judgment of the investigator, abnormal laboratory value of renal or hepatic function is clinically significant
* Known current (3 months prior to screening) or past (1 year prior to screening) abuse of alcohol or drugs, and/or current or past smoking habit of more than 10 cigarettes per day
* Any known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the trial with the exception of controlled thyroid function disease
* Known history of chemotherapy (except for gestational conditions) or radiotherapy
* According to the judgment of the investigator, abnormal laboratory value is clinically relevant
* Use of any non-registered investigational drugs during 3 months before screening or previous participation in the study

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 263 (Actual)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The number of retrieved oocytes per cycle | About 36 hours post hCG (human chorionic gonadotrophin)

SECONDARY OUTCOMES:
The follicles development | At day 5 of FSH preparation stimulation and the day of hCG administration
The fertilization rate | 20h (± 1h) after insemination
Implantation rate | 5-6 weeks post embryo transfer
Cycle cancellation rate | 36 hours post hCG
The positive serum β-hCG/hCG rate | 13-15 days after embryo transfer
The clinical pregnancy rate | 5-6 weeks after embryo transfer
  Regardless of fetal heart beat
The clinical pregnancy rate | 5-6 weeks after embryo transfer
  With fetal heart beat
The ongoing pregnancy rate | 10-11 weeks after embryo transfer
Total gonadotropin dose administered and the duration of gonadotropin treatment | Up to day 16 (in the stimulation period)
Serum E2 (Estradiol) concentrations | On the day of hCG administration
Frequency and severity of adverse events | Expected maximum of 7 months
Frequency and severity of injection site reactions | Day 1 up to day 16 of the controlled ovarian stimulation period
  Injection site reactions (in terms of "redness", "pain", "itching", "swelling" and "bruising")

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (11):
- China (11):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - The third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Tongji Hospital Tongji Medical College of HUST Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality